CLINICAL TRIAL: NCT01313689
Title: An Open Label, Multicenter Study Investigating the Safety and Efficacy of Ofatumumab Therapy Versus Physicians' Choice in Patients With Bulky Fludarabine-Refractory Chronic Lymphocytic Leukaemia (CLL)
Brief Title: Ofatumumab vs Physician's Choice in Subjects With Bulky Fludarabine-Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 114242
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Leukaemia
Keywords: OMB157; Lymphocytic; Chronic; Safety; Refractory; Chronic Lymphocytic Leukemia; Oncology; Ofatumumab; Efficacy; Physicians' Choice; Bulky Fludarabine Refractory Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia; Bronchiolitis Obliterans Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ofatumumab (Experimental): Biological
  Interventions: Drug: Ofatumumab
- Physicians' Choice (Active Comparator): Physicians' choice of treatment
  Interventions: Drug: Physicians' Choice

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab IV, initial dose 300 mg, followed 1 week later with 2000 mg once weekly for 7 weeks, followed 4 weeks later by one infusion of 2000 mg every 4 weeks for 4 infusions, for a total of 12 infusions over 24 weeks. After 24 weeks of ofatumumab treatment, patients who have achieved at least stable disease or better, and whom the investigator would deem appropriate for the therapy to continue, would undergo a second randomisation (2:1) to either 1) an additional ofatumumab dose regimen of 2000 mg once every 4 weeks for up to an additional 24 weeks, or 2) no further therapy (i.e. observation only).
  Arms: Ofatumumab
Drug: Physicians' Choice — Non-ofatumumab containing regimen as per physicians' choice for up to 6 months. Permitted therapies include treatments approved for CLL, and well established standards of care for CLL.
  Arms: Physicians' Choice

SUMMARY:
The purpose of this study was to confirm the clinical benefit observed in the pivotal registration study, Hx-CD20-406. The Committee for Medicinal Products for Human Use (CHMP) required that a randomized study be conducted in CLL patients with bulky fludarabine-refractory disease as a specific obligation for grant of conditional approval for ARZERRA™ in the European Union (EU). This study compared ofatumumab with the physicians' choice of therapy.

DETAILED DESCRIPTION:
Patients with CLL that is refractory to fludarabine have few treatment options and a poor prognosis. There is a continued need for new therapies for these CLL patients, as demonstrated by the limited responses and substantial toxicities with existing therapies. This is supported by the lack of a consensus around standard of care treatment for CLL patients with bulky fludarabine-refractory disease. The objective of this study was to confirm the response rate and disease control in the refractory setting through a controlled trial comparing ofatumumab with the physicians' choice of therapy in fludarabine-refractory, bulky lymphadenopathy patients. After 24 weeks of treatment with ofatumumab, patients were further randomized to either extended ofatumumab treatment or observation. Patients on the physicians' choice arm had the option of receiving ofatumumab if they experience progressive disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults with documented diagnosis of active CLL requiring treatment
* Bulky lymphadenopathy, defined as at least 1 lymph node >5 cm
* Must be refractory to fludarabine treatment
* Age 18 yrs or older
* At least 2 prior therapies for CLL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Signed written informed consent

Exclusion Criteria:

* Prior allogeneic stem cell transplant at any time, or autologous stem cell transplant within 6 months
* Treatment with any unapproved drug substance or experimental therapy within 4 weeks, or currently participating in another interventional clinical study
* CLL transformation, prolymphocytic leukemia, or central nervous system (CNS) involvement of CLL
* Active autoimmune hemolytic anemia (AIHA) requiring treatment except if associated with progressive disease requiring anti-CLL treatment
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment
* Human immunodeficiency virus (HIV) positive
* Significant concurrent, uncontrolled medical condition
* Other past or current malignancy (with the exception of basal cell carcinoma of the skin or in situ carcinoma of the cervix or breast) unless the tumor was successfully treated with curative intent at least 2 years prior to trial entry
* Non-protocol corticosteroid usage except a maintenance dose corresponding to less than or equal to 10 mg prednisone
* Abnormal lab values: Creatinine > 2.0 times upper normal limit (unless normal creatinine clearance), or total bilirubin > 2.0 times upper normal limit (unless due to liver involvement of CLL or due to Gilbert's syndrome), or alanine transaminase (ALT) > 2.5 times upper normal limit (unless due to liver involvement of CLL)
* Known or suspected hypersensitivity to ofatumumab
* Lactating or pregnant women or female patients of child-bearing potential (or male patients with such partners) not willing to use adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2014-03-18 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (75):
- Austria (5):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Novartis Investigative Site, Sofia, Bulgaria
- Czechia (3):
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (8):
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
- Germany (10):
  - Novartis Investigative Site, Kronach, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Frankfurt (Oder), Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Koblenz, Rhineland-Palatinate
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szombathely
- Ireland (3):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
  - Novartis Investigative Site, James Street
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (5):
  - Novartis Investigative Site, Modena, Emilia-Romagna
  - Novartis Investigative Site, Brescia, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Turin, Piedmont
  - Novartis Investigative Site, Messina, Sicily
- Poland (3):
  - Novartis Investigative Site, Chorzów
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Wroclaw
- Russia (4):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, St'Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Slovakia (3):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Martin
- Sweden (7):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Ukraine (11):
  - Novartis Investigative Site, Cherkasy
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Kharkiv
  - Novartis Investigative Site, Khmelnytskyi
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Makiivka
  - Novartis Investigative Site, Simferopil
  - Novartis Investigative Site, Vinnitsa
  - Novartis Investigative Site, Zhytomyr
- United Kingdom (3):
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Osterborg A, Udvardy M, Zaritskey A, Andersson PO, Grosicki S, Mazur G, Kaplan P, Steurer M, Schuh A, Montillo M, Kryachok I, Middeke JM, Kulyaba Y, Rekhtman G, Gorczyca M, Daly S, Chang CN, Lisby S, Gupta I. Phase III, randomized study of ofatumumab versus physicians' choice of therapy and standard versus extended-length ofatumumab in patients with bulky fludarabine-refractory chronic lymphocytic leukemia. Leuk Lymphoma. 2016 Sep;57(9):2037-46. doi: 10.3109/10428194.2015.1122783. Epub 2016 Jan 19. PMID 26784000

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: The 'Total Participants' in the Baseline Characteristics Table and in most of the Efficacy results Tables should be either Any OFA + Physician's Choice or OFA extended + OFA observation + OFA + Physician's Choice instead of the automatic calculated Total number indicated.
Pre-assignment Details: Participants(par) were randomized to receive an Open-Label treatment(trt) of ofatumumab(OFA) or a physicians choice(PC) trt for up to 24 weeks. OFA par without progressive disease(PD) underwent a second randomization to receive an additional 24 weeks of OFA or no further trt. PC par who developed PD had the option to receive OFA salvage therapy.
Groups:
- Any Ofatumumab: Participants (par.) were randomized to receive ofatumumab (OFA) at Randomization 1. Par. were initially administered OFA 300 milligrams (mg) intravenously (IV). Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Following Randomization 1, par. not demonstrating PD entered Randomization 2 (OFA Extended or OFA Observation); or par. entered Survival Follow-up (SFU) if demonstrating progressive disease (PD). During Randomization 2, par. either received another 24 weeks of OFA 2000 mg every 4 weeks (OFA Extension) or received no further treatment (trt) (OFA Observation). Par. entered Follow-up until withdrawal or the end of study (60 months). Par only entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Physician's Choice (PC): Par. randomized to receive PC trt during Randomization 1 were admin. treatments approved for Chronic Lymphocytic Leukaemia (CLL) & well-established standards of care as prescribed with standard dose & route. Experimental therapies or any doses beyond approved/standard of care dose ranges were not allowed. Par. who developed PD during PC trt or Follow-up had the option to receive (single-agent) OFA salvage trt. Par. received an initial IV dose of OFA 300 mg. One week later, par. received OFA 2000 mg followed by 7 weekly infusions of OFA 2000 mg, followed by infusions of OFA 2000 mg every 4 weeks until Week 48, for max. trt duration of 48 weeks. Par. entered Follow-up after OFA salvage trt until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during OFA salvage trt. Only the survival status & anti-cancer therapy information was collected in the SFU. Par. did not receive OFA salvage trt & demonstrated PD, entered SFU.Of 43 par 22 went to OFA salvage arm.
- Ofatumumab Extended (OFA Ext): Par. randomized to receive OFA at Randomization 1 and at Randomization 2. Only the par. who did not demonstrate PD during the first 24 weeks of OFA therapy entered Randomization 2. At Randomization 1, par. were initially administered OFA 300 mg IV. Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Par. randomized to Randomization 2 continued to receive OFA 2000 mg IV every 4 weeks for another 24 weeks. Par. entered Follow-up after the treatment period until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Ofatumumab Observation (OFA Observ.): Par. randomized to receive OFA at Randomization 1 and receiving no treatment at Randomization 2. Only the par. who did not demonstrate PD during the first 24 weeks of OFA therapy entered Randomization 2. At Randomization 1, par. were initially administered OFA 300 mg IV. Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Par. randomized to Randomization 2 received no treatment for another 24 weeks. Par. entered Follow-up after the treatment period until withdrawal or at end of study (60 months). Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- OFA First Randomization Only (OFA FRO): Participants (par.) were randomized to receive ofatumumab (OFA) at Randomization 1. Par. were initially administered OFA 300 milligrams (mg) intravenously (IV). Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. These participants were only randomized once and did not get make it to the second randomization.
  Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
Period: 24-Week Randomization 1
Arm/Group | Any Ofatumumab | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO)
Started | 79 | 43 (Of the 43 participants in the PC arm, 22 entered the OFA Salvage arm.) | 0 | 0 | 0
Completed | 60 (Par. not entering Randomization 2 continued visits for Follow-up and overall survival assessment) | 33 (Par. that did not receive OFA salvage continued visits for Follow-up and overall survival assessment) | 0 | 0 | 0
Not Completed | 19 | 10 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 0 | 0 | 0
Period: 24-Week Randomization 2
Arm/Group | Any Ofatumumab | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO)
Started | 0 | 0 | 24 (Not all participants from Randomization 1 continued to Randomization 2.) | 13 (Not all participants from Randomization 1 continued to Randomization 2.) | 42 (OFA Participants who did not enter Randomization 2.)
Completed | 0 | 0 | 21 | 12 | 27
Not Completed | 0 | 0 | 3 | 1 | 15
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included subjects who were randomized. Note: The Total participants in the Baseline Characteristics Table & in most of the Efficacy results Tables should be either Any OFA + Physician's Choice or OFA extended + OFA observation + OFA + Physician's Choice instead of the automatic calculated Total number indicated
Groups:
- Any Ofatumumab (OFA): Participants (par.) were randomized to receive ofatumumab (OFA) at Randomization 1. Par. were initially administered OFA 300 milligrams (mg) intravenously (IV). Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Following Randomization 1, par. not demonstrating PD entered Randomization 2 (OFA Extended or OFA Observation); or par. entered Survival Follow-up (SFU) if demonstrating progressive disease (PD). During Randomization 2, par. either received another 24 weeks of OFA 2000 mg every 4 weeks (OFA Extension) or received no further treatment (trt) (OFA Observation). Par. entered Follow-up until withdrawal or the end of study (60 months). Par only entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Total: Total of all reporting groups
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO) | Total
Number analyzed (Participants) | 79 | 43 | 24 | 13 | 42 | 201
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The Intent-to-Treat (ITT) population included subjects who were randomized.
  Years | 63.3 (8.95) | 61.8 (9.87) | 61.7 (9.09) | 66.7 (5.99) | 63.2 (9.52) | 62.8 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Intent-to-Treat (ITT) population included subjects who were randomized.
  Participants
    Female | 24 | 14 | 9 | 2 | 13 | 62
    Male | 55 | 29 | 15 | 11 | 29 | 139
Race/Ethnicity, Customized [Number; unit: Participants] — Population: The Intent-to-Treat (ITT) population included subjects who were randomized.
  Participants
    Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
    Not Hispanic or Latino | 78 | 43 | 24 | 13 | 41 | 199

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Independent Review Committee (IRC)
Description: PFS is the interval of time between the date of first randomization to the date of disease progression (PD) or death due to any reason, whichever occurred first. The date of PD was defined as the first occurrence of any criteria of progression. PD criteria requires at least one of the following: progression of lymphadenopathy, >=50% increase in liver or spleen size, >=50% increase in number of lymphocytes per microliter, more aggressive histology, occurence of cytopenia after treatment attributable to CLL. Disease progression was determined according to the 2008 International Workshop for Chronic Lymphocytic Leukaemia (IWCLL) update of the National Cancer Institute-sponsored Working Group CLL Guidelines for Response (NCI-WG). PFS was censored at the time of the last follow up for participants who have neither progressed or died.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: Intent-to-treat (ITT) population: all participants who were randomised to receive OFA or PC at the first randomisation.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ofatumumab Observation (OFA Observ.): These participants came from the Physicia's Choice (PC) arm. Par. randomized to receive OFA at Randomization 1 and receiving no treatment at Randomization 2. Only the par. who did not demonstrate PD during the first 24 weeks of OFA therapy entered Randomization 2. At Randomization 1, par. were initially administered OFA 300 mg IV. Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Par. randomized to Randomization 2 received no treatment for another 24 weeks. Par. entered Follow-up after the treatment period until withdrawal or at end of study (60 months). Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 79 | 43 | 24 | 13
Months | 5.36 [4.30 to 6.97] | 3.61 [1.87 to 6.74] | 10.05 [7.23 to 13.80] | 7.16 [5.36 to 9.49]
Statistical Analysis 1: Comparison: Any Ofatumumab (OFA) vs Physician's Choice (PC); Test type: Superiority or Other; p = 0.2677, Log Rank; P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.50 to 1.24] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum
Statistical Analysis 2: Comparison: Ofatumumab Extended (OFA Ext) vs Ofatumumab Observation (OFA Observ.); Test type: Superiority or Other; p = 0.0837, Log Rank; P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.19 to 1.53] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum

2. Secondary Outcome: Progression-free Survival (PFS) as Assessed by Investigator
Description: as for outcome 1
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: Intent-to-treat (ITT) population: all participants who were randomised to receive OFA or PC at the first randomisation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 79 | 43 | 24 | 13
Months | 7.00 [5.42 to 8.25] | 4.50 [1.97 to 5.62] | 12.68 [10.09 to 14.29] | 9.49 [7.00 to 12.12]
Statistical Analysis 1: Comparison: Any Ofatumumab (OFA) vs Physician's Choice (PC); Test type: Superiority or Other; p = 0.0030, Log Rank; P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.35 to 0.87] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum
Statistical Analysis 2: Comparison: Ofatumumab Extended (OFA Ext) vs Ofatumumab Observation (OFA Observ.); Test type: Superiority or Other; p = 0.0262, Log Rank; P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.21 to 1.17] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum

3. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the IRC
Description: ORR is defined as the number of participants achieving either complete response (CR) or partial response (PR). ORR was measured using the IWCLL updated NCI-WG guidelines 2008. CR requires all of the following criteria: no lymphadenopathy(Ly)/ hepatomegaly, splenomegaly, constitutional symptoms; neutrophils >1500 per microliter(µL), platelets(PL) >100,000/µL, hemoglobin(Hb) >11 grams/deciliter(g/dL), lymphocytes(LC) <4000/µL, bone marrow(BM) sample must be normocellular for age, <30% LC and no lymphoid nodules. PR requires the following criteria for at least 2 months: >=50% decrease in LC, reduction in Ly (i.e., >=50% decrease in lymph node size or no increase or new lymph nodes), >=50% decrease in the size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline(BL), Hb >11 g/dL or 50% improvement over BL, neutrophils>1500/μL. Nodular PR (nPR) indicates persistent nodules in the BM.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT Population. Not evaluable is defined as insufficient data present to classify into one of the other categories.
Measure: Number; unit: Participants
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 79 | 43 | 24 | 13
Participants
  CR | 0 | 0 | 0 | 0
  PR | 30 | 7 | 18 | 8
  nPR | 0 | 0 | 0 | 0
  Stable Disease | 36 | 22 | 5 | 5
  Progressive Disease | 9 | 8 | 1 | 0
  Not Evaluable | 4 | 6 | 0 | 0
  Missing | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Any Ofatumumab (OFA) vs Physician's Choice (PC); Test type: Superiority or Other; p = 0.0223, Regression, Logistic; conditional logistic regression with interval and pooled stratum; Odds Ratio (OR) = 2.942, 95% CI 2-sided [1.166 to 7.424]
Statistical Analysis 2: Comparison: Ofatumumab Extended (OFA Ext) vs Ofatumumab Observation (OFA Observ.); Test type: Superiority or Other; p = 0.9985, Regression, Logistic; conditional logistic regression with interval and pooled stratum; Odds Ratio (OR) = 999.999, 95% CI 2-sided [0.001 to 999.999]

4. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator
Description: ORR is defined as the number of participants achieving either complete response (CR) or partial response (PR). Overall response was measured using the IWCLL updated NCI-WG guidelines 2008. CR requires all of the following criteria: no lymphadenopathy(Ly)/ hepatomegaly, splenomegaly, constitutional symptoms; neutrophils >1500 per microliter(µL), platelets(PL) >100,000/µL, hemoglobin(Hb) >11 grams/deciliter(g/dL), lymphocytes(LC) <4000/µL, bone marrow(BM) sample must be normocellular for age, <30% LC and no lymphoid nodules. PR requires the following criteria for at least 2 months: >=50% decrease in LC, reduction in Ly (i.e., >=50% decrease in lymph node size or no increase or new lymph nodes), >=50% decrease in the size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline(BL), Hb >11 g/dL or 50% improvement over BL, neutrophils>1500/μL. Nodular PR (nPR) indicates persistent nodules in the BM.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT Population. Not evaluable is defined as insufficient data present to classify into one of the other categories.
Measure: Number; unit: Participants
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO)
Number analyzed (Participants) | 79 | 43 | 24 | 13 | 42
Participants
  CR | 2 | 2 | 1 | 1 | 0
  PR | 36 | 12 | 17 | 7 | 12
  nPR | 1 | 2 | 0 | 1 | 0
  Stable Disease | 34 | 14 | 6 | 4 | 24
  Progressive Disease | 2 | 10 | 0 | 0 | 2
  Not Evaluable | 0 | 0 | 0 | 0 | 0
  Missing | 4 | 3 | 0 | 0 | 4
Statistical Analysis 1: Comparison: Any Ofatumumab (OFA) vs Physician's Choice (PC); Test type: Superiority or Other; p = 0.4159, Regression, Logistic — Odds ratios and p-value are based on conditional logistic regression with interval and pooled stratum included in the Strata statement; Odds Ratio (OR) = 1.366, 95% CI 2-sided [0.644 to 2.899]
Statistical Analysis 2: Comparison: Ofatumumab Extended (OFA Ext) vs Ofatumumab Observation (OFA Observ.); Test type: Superiority or Other; p = 0.8866, Regression, Logistic — Odds ratios and p-value are based on conditional logistic regression with interval and pooled stratum in the strata statement; Odds Ratio (OR) = 1.225, 95% CI 2-sided [0.076 to 19.862]

5. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from randomization to death due to any cause. Kaplan-Meier plots were used to estimate the reported median OS time.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT population. Only those participants with data available were analyzed, participants who had not died were censored at the date of last contact.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO)
Number analyzed (Participants) | 79 | 43 | 24 | 13 | 42
Months | 19.19 [12.19 to 29.11] | 14.52 [8.94 to 24.97] | 31.54 [19.19 to 51.25] | 45.50 [14.69 to NA] — N/A = The upper limit of the 95% CI is not available due to the sparcity of the data. | 8.57 [4.93 to 16.76]
Statistical Analysis 1: Comparison: Any Ofatumumab (OFA) vs Physician's Choice (PC); Test type: Superiority or Other; p = 0.1732, Log Rank; P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.48 to 1.17] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum
Statistical Analysis 2: Comparison: Ofatumumab Extended (OFA Ext) vs Ofatumumab Observation (OFA Observ.); Test type: Superiority or Other; p = 0.8128, Log Rank — P-value is based on the stratified log-rank test adjusted for 'interval' and pooled stratum; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.46 to 2.68] — Hazard ratios are estimated using the Pike estimator, adjusted for 'interval' and pooled stratum

6. Secondary Outcome: Time to Progression as Assessed by IRC
Description: Time to progression is defined as the time from the date of randomization to disease progression (PD). PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlarged lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Participants who were alive and had not progressed at the time of analysis or if a progression event occurred after extensive lost-to-follow-up time were censored at the date of the last visit with adequate assessment.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT population. Only those participants with data available were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 56 | 23 | 19 | 11
Months | 6.31 [4.83 to 7.33] | 5.32 [2.14 to 8.08] | 10.05 [7.23 to 13.80] | 7.16 [5.36 to 9.49]

7. Secondary Outcome: Time to Next Anti-cancer Therapy by Investigator
Description: Time to next therapy is defined as the time from randomization until the start of the next line of treatment.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT population. Only those participants with data available were analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 44 | 29 | 12 | 12
Months | 11.50 [8.51 to 13.80] | 6.54 [2.66 to 8.08] | 15.47 [11.86 to NA] — The upper limit of the 95% CI is not available due to the sparcity of the data. | 9.00 [8.08 to 14.16]

8. Secondary Outcome: Time to Response as Assessed by the IRC
Description: Time to response is defined as the time from randomization to the first response (Complete Remission[CR], Complete Remission with incomplete bone marrow recovery[CRi], partial response[PR], or nodular PR[nPR]). CR(all the criteria at least 2 months after last treatment): no lymphadenopathy(Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter(µL), platelets(PL) >100,000/µL, hemoglobin(Hb) >11 grams/deciliter(g/dL), lymphocytes(LC) <4000/µL, bone marrow(BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline(BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM. Participants with unknown or missing responses were considered as non-responders.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT population. Only responders (CR, CRi, PR, nPR) were included in the analysis. Response was measured using the International Workshop for CLL (IWCLL) updated National Cancer Institute-sponsored Working Group (NCI-WG) guidelines 2008.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 30 | 7 | 18 | 8
Months | 1.17 [1.02 to 1.91] | 2.56 [0.76 to 3.48] | 1.86 [1.05 to 1.94] | 1.15 [0.92 to 1.94]

9. Secondary Outcome: Duration of Response as Assessed by the IRC
Description: DOR is defined as the time from the initial response (CR, CRi, nPR, or PR) to the first documented sign of PD or death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlarged lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Par. who were alive and had not progressed at the time of analysis or if a progression event occurred after extensive lost-to-follow-up time (>= 12 weeks) were censored at the date of the last visit with adequate assessment. Par. with unknown or missing responses were considered as non-responders.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: ITT population. Only those participants with data available at the indicated time points were analyzed. Only responders (CR, CRi, PR, nPR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC)
Number analyzed (Participants) | 23 | 5
Months | 6.24 [5.32 to 12.22] | 6.95 [4.47 to NA] — The upper limit of the 95% CI is not available due to the sparcity of the data.

10. Secondary Outcome: Number of Participants With Any Adverse Event (AE), Any Serious Adverse Event (SAE), Any Fatal Serious Adverse Event (FSAE), or Deaths
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability or incapacity, is a congenital anomaly or birth defect.
Time Frame: From the first dose of study medication to 60 days after the last dose of study medication and until follow-up for SAEs unless initiation of subsequent anti-CLL therapy
Population: Safety Population: all participants who received at least one dose of any study treatment (OFA or PC) at the first randomization.
Measure: Number; unit: Participants
Groups:
- OFA Salvage: The participants in this arm are from the Physician's Choice (PC) arm. Par. who developed PD during PC trt or Follow-up had the option to receive (single-agent) OFA salvage trt. Par. received an initial IV dose of OFA 300 mg. One week later, par. received OFA 2000 mg followed by 7 weekly infusions of OFA 2000 mg, followed by infusions of OFA 2000 mg every 4 weeks until Week 48, for the maximum trt duration of 48 weeks. Par. entered Follow-up after the OFA salvage trt until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during OFA salvage trt. Only the survival status and anti-cancer therapy information was collected in the SFU.
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO) | OFA Salvage
Number analyzed (Participants) | 78 | 43 | 24 | 13 | 41 | 22
Participants
  Any AE | 71 | 37 | 22 | 10 | 39 | 20
  Any SAE | 43 | 23 | 12 | 5 | 26 | 10
  Any FSAE | 14 | 6 | 2 | 3 | 9 | 5
  Deaths | 1 | 0 | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With Any Adverse Event (AE) of Special Interest
Description: AEs of special interest included cytopenias (neutropenia [decreased neutrophil count], anaemia [decreased hemoglobin], and thrombocytopenia [decreased platelet count]), autoimmune haematologic complications (autoimmune haemolytic anaemia and haemolytic anaemia), infusion reactions, infections, mucocutaneous reactions, Tumour Lysis Syndrome (TLS), cardiovascular events, and small bowel obstruction.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 78 | 43 | 24 | 13
Participants
  Any AE of decreased neutrophil count | 23 | 15 | 11 | 2
  Any AE of decreased hemoglobin | 9 | 9 | 3 | 2
  Any AE of decreased platelet count | 10 | 5 | 3 | 1
  Any AE of autoimmune haemolytic anaemia | 0 | 2 | 0 | 0
  Any AE of haemolytic anaemia | 1 | 0 | 1 | 0
  Any infusion related AE | 33 | 11 | 8 | 4
  Any AE of Infection | 46 | 24 | 16 | 8
  Any AE of mucocutaneous reaction | 20 | 4 | 6 | 3
  Any AE of TLS | 1 | 1 | 0 | 0
  Any AE of cardiovascular events | 13 | 3 | 6 | 0
  Any AE of small bowel obstruction | 0 | 0 | 0 | 0

12. Secondary Outcome: Mean Immunoglobulin (Ig) Antibodies IgA, IgG, and IgM Over Time
Description: Immunoglobulins or antibodies are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants. Immunoglobulin testing was performed at Screening (SCR), Cycle 3 Week 4 (C3W4), Cycle 7 Week 4 (C3W4) ,Cycle 9 Week 4 (C3W4), 6 Month Follow-up Visit (6M FU), 9 Month Follow-up (9M FU), 12 Month Follow-up (12M FU), 18 Month Follow-up (18M FU), 24 Month Follow-up (24M FU), 30 Month Follow-up (30M FU), 36 Month Follow-up (36M FU), 42 Month Follow-up (42M FU). A cycle is defined as the time between one round of treatment until the start of the next round.
Time Frame: Screening and every 3 months during treatment, every 6 months after last treatment until PD or until 42 Month Follow-up Visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Gram per liter
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO) | OFA Salvage
Number analyzed (Participants) | 78 | 43 | 24 | 13 | 41 | 22
Gram per liter
  IgA, SCR: number analyzed (Participants) | 78 | 41 | 24 | 13 | 41 | 0
  IgA, SCR | 0.793 (0.6680) | 0.685 (0.5518) | 0.807 (0.7426) | 1.095 (0.7535) | 0.688 (0.5749) |
  IgG, SCR: number analyzed (Participants) | 78 | 41 | 24 | 13 | 41 | 0
  IgG, SCR | 6.909 (4.6836) | 8.615 (12.1625) | 6.270 (3.8573) | 8.128 (4.7569) | 6.898 (5.1142) |
  IgM, SCR: number analyzed (Participants) | 77 | 41 | 24 | 13 | 40 | 0
  IgM, SCR | 0.800 (1.3154) | 0.601 (0.7061) | 0.800 (1.6649) | 0.468 (0.3801) | 0.907 (1.2822) |
  IgA, C3W4: number analyzed (Participants) | 61 | 23 | 24 | 12 | 25 | 17
  IgA, C3W4 | 0.721 (0.6355) | 0.675 (0.4819) | 0.808 (0.7931) | 0.977 (0.6458) | 0.514 (0.3621) | 0.486 (0.3868)
  IgG, C3W4: number analyzed (Participants) | 61 | 23 | 24 | 12 | 25 | 17
  IgG, C3W4 | 5.925 (3.5059) | 5.481 (2.1226) | 5.949 (3.4089) | 7.232 (4.0103) | 5.276 (3.3056) | 5.974 (2.7992)
  IgM, C3W4: number analyzed (Participants) | 61 | 23 | 24 | 12 | 25 | 17
  IgM, C3W4 | 0.692 (1.3420) | 0.485 (0.4929) | 0.882 (1.9833) | 0.429 (0.3497) | 0.636 (0.7764) | 0.488 (0.4816)
  IgA, C7W4: number analyzed (Participants) | 38 | 0 | 24 | 12 | 2 | 10
  IgA, C7W4 | 0.793 (0.6608) |  | 0.723 (0.6730) | 0.945 (0.6724) | 0.725 (0.6011) | 0.537 (0.4356)
  IgG, C7W4: number analyzed (Participants) | 38 | 0 | 24 | 10 | 2 | 10
  IgG, C7W4 | 6.250 (3.5225) |  | 5.817 (3.4944) | 7.254 (3.7588) | 5.420 (2.2062) | 5.135 (2.6309)
  IgM, C7W4: number analyzed (Participants) | 38 | 0 | 24 | 12 | 2 | 10
  IgM, C7W4 | 0.762 (1.7523) |  | 0.844 (2.1136) | 0.414 (0.3400) | 1.865 (2.3547) | 0.447 (0.4732)
  IgA, C9W4: number analyzed (Participants) | 29 | 0 | 21 | 8 | 0 | 7
  IgA, C9W4 | 0.719 (0.6336) |  | 0.630 (0.6005) | 0.952 (0.6997) |  | 0.567 (0.3968)
  IgG, C9W4: number analyzed (Participants) | 29 | 0 | 21 | 8 | 0 | 7
  IgG, C9W4 | 6.164 (3.5886) |  | 5.553 (3.0792) | 7.768 (4.5126) |  | 5.709 (2.1629)
  IgM, C9W4: number analyzed (Participants) | 29 | 0 | 21 | 8 | 0 | 7
  IgM, C9W4 | 0.853 (2.3484) |  | 0.973 (2.7574) | 0.536 (0.4209) |  | 0.484 (0.4493)
  IgA, 6M FU: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  IgA, 6M FU |  | 0.880 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |  |
  IgG, 6M FU: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  IgG, 6M FU |  | 8.670 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |  |
  IgM, 6M FU: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  IgM, 6M FU |  | 0.200 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |  |
  IgA, 9M FU: number analyzed (Participants) | 2 | 5 | 2 | 0 | 0 | 0
  IgA, 9M FU | 0.890 (0.0849) | 0.510 (0.4585) | 0.890 (0.0849) |  |  |
  IgG, 9M FU: number analyzed (Participants) | 2 | 5 | 2 | 0 | 0 | 0
  IgG, 9M FU | 7.695 (0.9263) | 5.016 (2.4292) | 7.695 (0.9263) |  |  |
  IgM, 9M FU: number analyzed (Participants) | 2 | 5 | 2 | 0 | 0 | 0
  IgM, 9M FU | 0.375 (0.1061) | 0.246 (0.0706) | 0.375 (0.1061) |  |  |
  IgA, 12M FU: number analyzed (Participants) | 10 | 3 | 7 | 3 | 0 | 2
  IgA, 12M FU | 0.721 (0.8339) | 0.983 (0.6029) | 0.826 (0.9960) | 0.477 (0.1595) |  | 0.300 (0.000)
  IgG, 12M FU: number analyzed (Participants) | 10 | 3 | 7 | 3 | 0 | 2
  IgG, 12M FU | 6.423 (3.5390) | 7.497 (1.5550) | 7.621 (3.3834) | 3.627 (2.2938) |  | 4.935 (0.8273)
  IgM, 12M FU: number analyzed (Participants) | 10 | 3 | 7 | 3 | 0 | 2
  IgM, 12M FU | 0.384 (0.3463) | 0.487 (0.2743) | 0.3334 (0.2833) | 0.500 (0.5197) |  | 0.240 (0.0566)
  IgA, 18M FU: number analyzed (Participants) | 8 | 2 | 7 | 1 | 0 | 2
  IgA, 18M FU | 0.520 (0.2803) | 1.095 (0.2616) | 0.500 (0.2965) | 0.660 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0.300 (0.000)
  IgG, 18M FU: number analyzed (Participants) | 8 | 2 | 7 | 1 | 0 | 2
  IgG, 18M FU | 4.513 (2.0789) | 6.620 (2.3759) | 4.206 (2.0405) | 6.660 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 4.265 (1.1384)
  IgM, 18M FU: number analyzed (Participants) | 8 | 2 | 7 | 1 | 0 | 2
  IgM, 18M FU | 0.417 (3.3156) | 0.640 (0.2687) | 0.317 (0.1490) | 1.120 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0.240 (0.0566)
  IgA, 24M FU: number analyzed (Participants) | 5 | 1 | 4 | 1 | 0 | 0
  IgA, 24M FU | 0.540 (0.2667) | 1.540 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.480 (0.2662) | 0.780 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  IgG, 24M FU: number analyzed (Participants) | 5 | 1 | 4 | 1 | 0 | 0
  IgG, 24M FU | 5.634 (2.4734) | 10.900 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 5.098 (2.4977) | 7.780 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  IgM, 24M FU: number analyzed (Participants) | 5 | 1 | 4 | 1 | 0 | 0
  IgM, 24M FU | 0.490 (0.3621) | 1.710 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.333 (0.0971) | 1.120 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  IgA, 30M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgA, 30M FU | 0.505 (0.2900) | 1.380 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.505 (0.2900) |  |  |
  IgG, 30M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgG, 30M FU | 3.460 (1.8809) | 11.100 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.460 (1.8809) |  |  |
  IgM, 30M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgM, 30M FU | 0.400 (0.1131) | 0.770 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.400 (0.1131) |  |  |
  IgA, 36M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgA, 36M FU | 0.550 (0.3111) | 1.680 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.550 (0.3111) |  |  |
  IgG, 36M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgG, 36M FU | 4.320 (2.2486) | 13.600 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 4.320 (2.2486) |  |  |
  IgM, 36M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgM, 36M FU | 1.175 (0.2899) | 0.720 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 1.175 (0.2899) |  |  |
  IgA, 42M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgA, 42M FU | 0.545 (0.2051) | 1.410 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0.545 (0.2051) |  |  |
  IgG, 42M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgG, 42M FU | 4.425 (3.5143) | 11.500 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 4.425 (3.5143) |  |  |
  IgM, 42M FU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  IgM, 42M FU | 2.155 (0.8697) | 0.470 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 2.155 (0.8697) |  |  |

13. Secondary Outcome: Number of Participants Who Were Positive or Negative for Human Anti-Human Antibodies (HAHA) Post-OFA Therapy
Description: The presence of HAHA in human serum was determined using a validated electrochemiluminescent assay in a multi-tier assay format. All samples were first assessed in a screening (SCR) assay, and the potential positive (Pos) samples were further tested in the confirmation (CNF) assays. Confirmed positives were reported as HAHA positive and titer was determined for each positive sample. The drug tolerance of the HAHA assay is 200 microgram/milliliter (µg/mL); thus, samples that tested negative in the assay and had ofatumumab concentrations no more than 200 µg/mL were considered as conclusive negative (Neg) results.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: Safety Population. Only those participants with post-OFA treatment HAHA results were analyzed.
Measure: Number; unit: Participants
Arm/Group | Any Ofatumumab (OFA) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO) | OFA Salvage
Number analyzed (Participants) | 78 | 24 | 13 | 41 | 22
Participants
  CNF Pos: number analyzed (Participants) | 69 | 24 | 13 | 32 | 19
  CNF Pos | 0 | 0 | 0 | 0 | 0
  Neg and no OFA concentration <200 ug/mL: number analyzed (Participants) | 69 | 24 | 13 | 32 | 19
  Neg and no OFA concentration <200 ug/mL | 12 | 1 | 1 | 10 | 4
  Neg and at least one OFA concentration <200 ug/mL: number analyzed (Participants) | 69 | 24 | 13 | 32 | 19
  Neg and at least one OFA concentration <200 ug/mL | 57 | 23 | 12 | 22 | 15

14. Secondary Outcome: Changes From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire, Chronic Lymphocytic Leukaemia 16 Item Module (EORTC QLQ-CLL 16)
Description: The EORTC QLQ-CLL16 is comprised of 16 questions that address 5 domains of health-related quality of life (HRQoL) important in CLL. There are 4 multi-item scales - fatigue (2 items), treatment side effects ([TSE], 4 items), disease symptoms (disease effects scale [DES], 4 items), and infection (4 items) - and single item scales (social activities [Social Problems (SP) Scale] and future health worries[Future Health (FH) Scale].). These are measured on a four point scale where 1 = not at all and 4 = very much. These scores are transformed to give a rating from 0 - 100, where 0 =no symptoms or problems and 100 = a severe symptoms or problems. EORTC QLQ-CLL16 was assessed at Screening; Week (W) 12 (W4 of Cycle[C] 3), W24 (W4C6), W36 (W4C9), W48 (W4C13); during Follow-up which was every month for Months (M) 1-6, every 8 weeks for M7-12 and every 3 months up to M60; and then at PD.
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: Intent-to-treat (ITT) population: all participants who were randomised to receive OFA or PC at the first randomisation.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.)
Number analyzed (Participants) | 79 | 43 | 24 | 13
unit on a scale
  DES, C3W4: number analyzed (Participants) | 59 | 21 | 24 | 12
  DES, C3W4 | -10.3 (17.60) | -6.3 (16.22) | -9.7 (12.20) | -10.4 (17.09)
  DES, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  DES, C6W4 | -8.5 (15.82) | -6.4 (16.37) | -8.3 (14.95) | -9.8 (18.19)
  DES, C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  DES, C9W4 | -11 (17.72) |  | -7.5 (17.91) | -19.8 (14.73)
  DES, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  DES, C12W4 | -3.3 (21.78) |  | -3.3 (21.78) |
  DES, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  DES, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  DES, 5MFU |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  DES, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  DES, 6MFU |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  DES, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  DES, 7MFU |  | -14.6 (16.52) |  |
  DES, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  DES, 9MFU | 0 (23.57) | -9.7 (9.74) | 0 (23.57) |
  DES, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  DES, 11MFU | -25 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -6.7 (18.07) | -25 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  DES, 12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  DES, 12MFU | -10.8 (14.19) | -2.8 (20.97) | -10.4 (14.6) | -12.5 (17.68)
  DES, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  DES, 15MFU | -4.8 (13.49) | -5.6 (17.35) | -4.8 (13.49) |
  DES, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  DES, 18MFU | -3.3 (13.94) | -20.8 (17.68) | -3.3 (13.94) |
  DES, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  DES, 21MFU | 5.6 (20.97) | -12.5 (5.89) | 5.6 (20.97) |
  DES, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  DES, 24MFU | 4.2 (5.89) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 4.2 (5.89) |
  DES, 27MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  DES, 27MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  DES, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  DES, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Fatigue Scale, C3W4: number analyzed (Participants) | 59 | 21 | 24 | 12
  Fatigue Scale, C3W4 | -4 (24.04) | 2.4 (21.91) | -2.1 (19.23) | -12.5 (24.75)
  Fatigue Scale, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  Fatigue Scale, C6W4 | -5.7 (19.99) | 12.8 (29.78) | -0.7 (16.65) | -13.6 (19.46)
  Fatigue Scale, C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  Fatigue Scale, C9W4 | -4.2 (25.1) |  | 0 (24.78) | -14.6 (24.3)
  Fatigue Scale, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  Fatigue Scale, C12W4 | 7.8 (33.85) |  | 7.8 (33.85) |
  Fatigue Scale, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  Fatigue Scale, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Fatigue Scale, 5MFU |  | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Fatigue Scale, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Fatigue Scale, 6MFU |  | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Fatigue Scale, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  Fatigue Scale, 7MFU |  | -14.6 (18.77) |  |
  Fatigue Scale, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  Fatigue Scale, 9MFU | 41.7 (82.5) | -8.3 (22.97) | 41.7 (82.5) |
  Fatigue Scale, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  Fatigue Scale, 11MFU | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -6.7 (19) | -16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Fatigue Scale,12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  Fatigue Scale,12MFU | 5 (20.86) | -22.2 (9.62) | 6.3 (21.71) | 0 (23.57)
  Fatigue Scale, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  Fatigue Scale, 15MFU | 2.4 (22.42) | 0 (16.67) | 2.4 (22.42) |
  Fatigue Scale, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  Fatigue Scale, 18MFU | 3.3 (21.73) | 0 (0) | 3.3 (21.73) |
  Fatigue Scale, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  Fatigue Scale, 21MFU | 16.7 (28.87) | 0 (23.57) | 16.7 (28.87) |
  Fatigue Scale, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  Fatigue Scale, 24MFU | 41.7 (58.93) | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 41.7 (58.93) |
  Fatigue Scale, 27MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Fatigue Scale, 27MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Fatigue Scale, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Fatigue Scale, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Future Health Scale, C3W4: number analyzed (Participants) | 58 | 21 | 24 | 11
  Future Health Scale, C3W4 | -6.9 (27.04) | -7.9 (31.46) | -4.2 (22.66) | -6.1 (29.13)
  Future Health Scale, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  Future Health Scale, C6W4 | -12.9 (29.83) | -5.1 (18.49) | -11.1 (25.38) | -24.2 (39.7)
  Future Health Scale, C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  Future Health Scale, C9W4 | -14.3 (27.86) |  | -11.7 (27.09) | -20.8 (30.54)
  Future Health Scale, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  Future Health Scale, C12W4 | -4.4 (39.57) |  | -4.4 (39.57) |
  Future Health Scale, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  Future Health Scale, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Future Health Scale, 5MFU |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Future Health Scale, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Future Health Scale, 6MFU |  | 33.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Future Health Scale, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  Future Health Scale, 7MFU |  | -12.5 (24.8) |  |
  Future Health Scale, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  Future Health Scale, 9MFU | 0 (47.14) | -22.2 (40.37) | 0 (47.14) |
  Future Health Scale, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  Future Health Scale, 11MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -13.3 (18.26) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Future Health Scale, 12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  Future Health Scale, 12MFU | -10 (31.62) | -11.1 (19.25) | -4.2 (33.03) | -33.3 (0)
  Future Health Scale, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  Future Health Scale, 15MFU | 19 (17.82) | -11.1 (19.25) | 19 (17.82) |
  Future Health Scale, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  Future Health Scale, 18MFU | 20 (18.26) | -16.7 (23.57) | 20 (18.26) |
  Future Health Scale, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  Future Health Scale, 21MFU | 22.2 (19.25) | -16.7 (23.57) | 22.2 (19.25) |
  Future Health Scale, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  Future Health Scale, 24MFU | 33.3 (47.14) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 33.3 (47.14) |
  Future Health Scale, 27MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Future Health Scale, 27MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Future Health Scale, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Future Health Scale, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Infection Scale, C3W4: number analyzed (Participants) | 59 | 21 | 24 | 12
  Infection Scale, C3W4 | 2.1 (23.6) | 3.2 (19.63) | -1 (20.01) | -5.6 (12.48)
  Infection Scale, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  Infection Scale, C6W4 | -3.7 (22.66) | 12.2 (25.6) | -5.6 (19.91) | -6.8 (19.3)
  Infection Scale,C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  Infection Scale,C9W4 | -7.4 (18.61) |  | -7.5 (16.86) | -7.3 (23.75)
  Infection Scale, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  Infection Scale, C12W4 | -11.7 (14.02) |  | -11.7 (14.02) |
  Infection Scale, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  Infection Scale, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Infection Scale, 5MFU |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Infection Scale, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  Infection Scale, 6MFU |  | 8.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  Infection Scale, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  Infection Scale, 7MFU |  | -9.4 (12.15) |  |
  Infection Scale, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  Infection Scale, 9MFU | 16.7 (23.57) | 0 (13.94) | 16.7 (23.57) |
  Infection Scale, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  Infection Scale, 11MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -6.7 (12.36) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Infection Scale, 12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  Infection Scale, 12MFU | -7.5 (20.58) | 2.8 (12.73) | -6.2 (20.29) | -12.5 (29.46)
  Infection Scale, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  Infection Scale, 15MFU | -2.4 (17.82) | -2.8 (20.97) | -2.4 (17.82) |
  Infection Scale, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  Infection Scale, 18MFU | 5 (12.64) | -8.3 (11.79) | 5 (12.64) |
  Infection Scale, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  Infection Scale, 21MFU | 2.8 (12.73) | 8.3 (0) | 2.8 (12.73) |
  Infection Scale, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  Infection Scale, 24MFU | 0 (0) | 8.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0 (0) |
  Infection Scale, 27MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Infection Scale, 27MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  Infection Scale, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  Infection Scale, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  SP Scale, C3W4: number analyzed (Participants) | 59 | 21 | 24 | 12
  SP Scale, C3W4 | -9 (27.56) | 3.2 (36.37) | -11.1 (23.4) | -13.9 (30.01)
  SP Scale, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  SP Scale, C6W4 | -10.6 (27.63) | 10.3 (31.58) | -9.7 (25.02) | -15.2 (31.14)
  SP Scale, C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  SP Scale, C9W4 | -13.1 (27.72) |  | -11.7 (29.17) | -16.7 (25.2)
  SP Scale, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  SP Scale, C12W4 | -11.1 (37.09) |  | -11.1 (37.09) |
  SP Scale, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  SP Scale, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  SP Scale, 5MFU |  | -33.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  SP Scale, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  SP Scale, 6MFU |  | -66.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  SP Scale, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  SP Scale, 7MFU |  | -16.7 (25.2) |  |
  SP Scale, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  SP Scale, 9MFU | 16.7 (70.71) | -5.6 (32.77) | 16.7 (70.71) |
  SP Scale, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  SP Scale, 11MFU | -33.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -6.7 (36.51) | -33.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  SP Scale, 12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  SP Scale, 12MFU | -16.7 (23.57) | -22.2 (19.25) | -16.7 (25.2) | -16.7 (23.57)
  SP Scale, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  SP Scale, 15MFU | -9.5 (37.09) | -11.1 (19.25) | -9.5 (37.09) |
  SP Scale, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  SP Scale, 18MFU | 0 (23.57) | -16.7 (23.57) | 0 (23.57) |
  SP Scale, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  SP Scale, 21MFU | -22.2 (38.49) | -16.7 (23.57) | -22.2 (38.49) |
  SP Scale, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  SP Scale, 24MFU | 33.3 (47.14) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 33.3 (47.14) |
  SP Scale, 27MFU: number analyzed (Participants) | 1 | 2 | 1 | 0
  SP Scale, 27MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | NA (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  SP Scale, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  SP Scale, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  TSE Scale, C3W4: number analyzed (Participants) | 59 | 21 | 24 | 12
  TSE Scale, C3W4 | -4.8 (15.33) | -1.5 (16.82) | -2.4 (10.85) | -8.3 (13.76)
  TSE Scale, C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11
  TSE Scale, C6W4 | -4.2 (14.33) | 3.2 (12.52) | -0.2 (11.32) | -9.1 (16.44)
  TSE Scale, C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8
  TSE Scale, C9W4 | -5.4 (15.75) |  | -3.7 (13.91) | -9.4 (20.14)
  TSE Scale, C12W4: number analyzed (Participants) | 15 | 0 | 15 | 0
  TSE Scale, C12W4 | -2.8 (14.66) |  | -2.8 (14.66) |
  TSE Scale, 3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0
  TSE Scale, 5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  TSE Scale, 5MFU |  | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  TSE Scale, 6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0
  TSE Scale, 6MFU |  | 16.7 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  TSE Scale, 7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0
  TSE Scale, 7MFU |  | -8.3 (17.82) |  |
  TSE Scale, 9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0
  TSE Scale, 9MFU | 8.3 (11.79) | -1.4 (9.74) | 8.3 (11.79) |
  TSE Scale, 11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0
  TSE Scale, 11MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | -1.7 (14.91) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  TSE Scale, 12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2
  TSE Scale, 12MFU | -4.2 (19.74) | 2.8 (12.73) | 0 (12.6) | -20.8 (41.25)
  TSE Scale, 15MFU: number analyzed (Participants) | 7 | 3 | 7 | 0
  TSE Scale, 15MFU | -8.3 (12.73) | 2.8 (9.62) | -8.3 (12.73) |
  TSE Scale, 18MFU: number analyzed (Participants) | 5 | 2 | 5 | 0
  TSE Scale, 18MFU | 6.7 (16.03) | 0 (11.79) | 6.7 (16.03) |
  TSE Scale, 21MFU: number analyzed (Participants) | 3 | 2 | 3 | 0
  TSE Scale, 21MFU | 8.3 (22.05) | 0 (0) | 8.3 (22.05) |
  TSE Scale, 24MFU: number analyzed (Participants) | 2 | 1 | 2 | 0
  TSE Scale, 24MFU | 4.2 (5.89) | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 4.2 (5.89) |
  TSE Scale, 27MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  TSE Scale, 27MFU | 8.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 8.3 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |
  TSE Scale, 30MFU: number analyzed (Participants) | 1 | 0 | 1 | 0
  TSE Scale, 30MFU | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |

15. Secondary Outcome: Mean Health Change Questionnaire (HCQ) Score
Description: The HCQ consists of a single question in which the participant is asked if he/she has experienced any change in his/her health overall since beginning the study. For HCQ, values from 1 to 9 were assigned to the 9 responses in the HCQ questionnaire, ranging from 1 for 'my health is a great deal better' to 9 for 'my health is a great deal worse' since the beginning of the study. A score of 3 or less indicates improvement from Baseline. HCQ was assessed at Screening; Week (W) 12 (W4 of Cycle[C] 3), W24 (W4C6), W36 (W4C9), W48 (W4C13); during follow-up which was every month for Months 1-6, every 8 weeks for M7-12 and every 3 months up to M60; and then at PD..
Time Frame: From the randomization date up to 60 months post the randomization date.
Population: Population Description:
  Intent-to-treat (ITT) population: all participants who were randomised to receive OFA or PC at the first randomisation.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Any Ofatumumab (OFA) | Physician's Choice (PC) | Ofatumumab Extended (OFA Ext) | Ofatumumab Observation (OFA Observ.) | OFA First Randomization Only (OFA FRO) | OFA Salvage
Number analyzed (Participants) | 79 | 43 | 24 | 13 | 42 | 22
Unit on a scale
  C3W4: number analyzed (Participants) | 60 | 21 | 24 | 12 | 24 | 17
  C3W4 | 2.8 (1.57) | 3.9 (2.01) | 2.5 (1.44) | 2.8 (0.97) | 3.2 (1.90) | 3.1 (1.92)
  C6W4: number analyzed (Participants) | 44 | 13 | 24 | 11 | 9 | 12
  C6W4 | 3.2 (2.04) | 3.5 (2.37) | 2.7 (1.66) | 2.9 (1.76) | 5.1 (2.37) | 3.0 (2.00)
  C9W4: number analyzed (Participants) | 28 | 0 | 20 | 8 | 0 | 7
  C9W4 | 2.8 (1.60) |  | 2.5 (1.36) | 3.5 (2.00) |  | 3.1 (2.48)
  C12W4: number analyzed (Participants) | 14 | 0 | 14 | 0 | 0 | 4
  C12W4 | 2.6 (1.99) |  | 2.6 (1.99) |  |  | 3.0 (1.83)
  3MFU: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  3MFU |  |  |  |  |  | 3.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation.
  5MFU: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  5MFU |  | 5.0 (NA) — No participants were analyzed for this category at this time point therefore there is no data to present. There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |  |
  6MFU: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0
  6MFU |  | 3.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |  |
  7MFU: number analyzed (Participants) | 0 | 8 | 0 | 0 | 0 | 0
  7MFU |  | 2.4 (1.30) |  |  |  |
  9MFU: number analyzed (Participants) | 2 | 6 | 2 | 0 | 0 | 0
  9MFU | 6.5 (2.12) | 3.5 (2.07) | 6.5 (2.12) |  |  |
  11MFU: number analyzed (Participants) | 1 | 5 | 1 | 0 | 0 | 0
  11MFU | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.0 (2.35) | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |
  12MFU: number analyzed (Participants) | 10 | 3 | 8 | 2 | 0 | 2
  12MFU | 3.4 (2.07) | 2.3 (1.53) | 3.5 (2.27) | 3.0 (1.41) |  | 2.0 (1.41)
  15MFU: number analyzed (Participants) | 10 | 3 | 9 | 1 | 0 | 3
  15MFU | 3.5 (2.27) | 3.7 (1.53) | 3.7 (2.35) | 2.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 2.0 (1.00)
  18MFU: number analyzed (Participants) | 7 | 2 | 6 | 1 | 0 | 2
  18MFU | 2.6 (2.15) | 4.5 (0.71) | 2.8 (2.23) | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  | 4.0 (4.24)
  21MFU: number analyzed (Participants) | 5 | 2 | 4 | 1 | 0 | 0
  21MFU | 2.0 (1.22) | 6.0 (1.41) | 2.3 (1.26) | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  24MFU: number analyzed (Participants) | 4 | 1 | 3 | 1 | 0 | 0
  24MFU | 2.5 (3.00) | 4.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.0 (3.46) | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  27MFU: number analyzed (Participants) | 3 | 1 | 2 | 1 | 0 | 0
  27MFU | 2.7 (2.89) | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.5 (3.54) | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |
  30MFU: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  30MFU | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |
  33MFU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  33MFU | 3.0 (2.83) | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.0 (2.83) |  |  |
  36MFU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  36MFU | 3.0 (2.83) | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.0 (2.83) |  |  |
  39MFU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  39MFU | 4.0 (4.24) | 7.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 4.0 (4.24) |  |  |
  42MFU: number analyzed (Participants) | 2 | 1 | 2 | 0 | 0 | 0
  42MFU | 3.0 (2.83) | 5.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 3.0 (2.83) |  |  |
  45MFU: number analyzed (Participants) | 1 | 1 | 1 | 0 | 0 | 0
  45MFU | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 7.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. | 1.0 (NA) — There were too few participants analyzed at this time point to calculate a standard deviation. |  |  |

ADVERSE EVENTS:
Time Frame: SAEs & AEs were collected from first dose of study medication to 60 days after last dose of study medication & until end of the follow-up period (60 months post the randomization date) for SAEs unless initiation of subsequent anti-CLL therapy. AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit
Groups:
- Ofatumumab Extended: Par. randomized to receive OFA at Randomization 1 and at Randomization 2. Only the par. who did not demonstrate PD during the first 24 weeks of OFA therapy entered Randomization 2. At Randomization 1, par. were initially administered OFA 300 mg IV. Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Par. randomized to Randomization 2 continued to receive OFA 2000 mg IV every 4 weeks for another 24 weeks. Par. entered Follow-up after the treatment period until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Ofatumumab Observation: Par. randomized to receive OFA at Randomization 1 and receiving no treatment at Randomization 2. Only the par. who did not demonstrate PD during the first 24 weeks of OFA therapy entered Randomization 2. At Randomization 1, par. were initially administered OFA 300 mg IV. Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. Par. randomized to Randomization 2 received no treatment for another 24 weeks. Par. entered Follow-up after the treatment period until withdrawal or at end of study (60 months). Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Ofatumumab: Participants (par.) were randomized to receive ofatumumab (OFA) at Randomization 1. Par. were initially administered OFA 300 milligrams (mg) intravenously (IV). Beginning at Week 2, par. were administered OFA 2000 mg once weekly for 7 weeks, followed by 4 infusions of OFA 2000 mg every 4 weeks for a total of 12 infusions over 24 weeks. These participants were only randomized once and did not get make it to the second randomization. Par. entered SFU if demonstrating PD during the study. Only the survival status and anti-cancer therapy information was collected in the SFU.
- Physicians Choice: Par. randomized to receive PC trt during Randomization 1 were administered treatments approved for Chronic Lymphocytic Leukaemia (CLL) and well established standards of care as prescribed with standard dose and route. Experimental therapies or any doses beyond the approved/standard of care dose ranges were not allowed. Par. who developed PD during PC trt or Follow-up had the option to receive s(ingleagent) OFA salvage trt. Par. received an initial IV dose of OFA 300 mg. One week later, par. received OFA 2000 mg followed by 7 weekly infusions of OFA 2000 mg, followed by infusions of OFA 2000 mg every 4 weeks until Week 48, for the maximum trt duration of 48 weeks. Par. entered Follow-up after the OFA salvage trt until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during OFA salvage trt. Only the survival status and anti-cancer therapy information was collected in the SFU. Par. who did not receive OFA salvage trt and demonstrated PD, entered SFU
- Ofatumumab Salvage: Par. who developed PD during PC trt or Follow-up had the option to receive (single-agent) OFA salvage trt. Par. received an initial IV dose of OFA 300 mg. One week later, par. received OFA 2000 mg followed by 7 weekly infusions of OFA 2000 mg, followed by infusions of OFA 2000 mg every 4 weeks until Week 48, for the maximum trt duration of 48 weeks. Par. entered Follow-up after the OFA salvage trt until withdrawal or the end of study (60 months). Par. entered SFU if demonstrating PD during OFA salvage trt. Only the survival status and anticancer therapy information was collected in the SFU.
Arm/Group | Any Ofatumumab | Ofatumumab Extended | Ofatumumab Observation | Ofatumumab | Physicians Choice | Ofatumumab Salvage
All-Cause Mortality (participants affected / at risk) | 16/78 | 2/24 | 3/13 | 11/41 | 8/43 | 5/22
Serious Adverse Events (participants affected / at risk) | 43/78 | 12/24 | 5/13 | 26/41 | 23/43 | 10/22
Other Adverse Events (participants affected / at risk) | 63/78 | 20/24 | 10/13 | 33/41 | 30/43 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Ofatumumab (N=78) | Ofatumumab Extended (N=24) | Ofatumumab Observation (N=13) | Ofatumumab (N=41) | Physicians Choice (N=43) | Ofatumumab Salvage (N=22)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 4 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 1 | 6 | 4 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 2 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0 | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 1 | 0 | 1 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 0 | 0 | 1 | 0 | 0
Chorioretinal atrophy (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 0 | 0 | 4 | 3 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal fungal infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Otosalpingitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 10 | 3 | 1 | 6 | 7 | 3
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 2
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Chorea (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 2 | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Ofatumumab (N=78) | Ofatumumab Extended (N=24) | Ofatumumab Observation (N=13) | Ofatumumab (N=41) | Physicians Choice (N=43) | Ofatumumab Salvage (N=22)
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 0 | 3 | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 15 | 10 | 1 | 4 | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 3 | 1 | 4 | 3 | 1
Cardiac failure (Cardiac disorders) | 3 | 2 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 2 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 0 | 5 | 4 | 2
Nausea (Gastrointestinal disorders) | 8 | 2 | 1 | 5 | 5 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0 | 4 | 3 | 0
Asthenia (General disorders) | 3 | 0 | 0 | 3 | 0 | 0
Chills (General disorders) | 9 | 1 | 2 | 6 | 1 | 0
Fatigue (General disorders) | 3 | 0 | 1 | 2 | 4 | 0
Oedema peripheral (General disorders) | 2 | 0 | 1 | 1 | 3 | 0
Peripheral swelling (General disorders) | 4 | 1 | 0 | 3 | 1 | 0
Pyrexia (General disorders) | 8 | 2 | 1 | 5 | 3 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 7 | 5 | 0 | 2 | 3 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 0
Eye infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 5 | 3 | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3 | 0 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 1 | 1 | 2 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 2 | 2 | 5 | 2
Urinary tract infection (Infections and infestations) | 3 | 0 | 0 | 3 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1 | 1 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 1 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 1 | 2 | 2
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 3 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 3 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 3 | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 2
Headache (Nervous system disorders) | 3 | 0 | 0 | 3 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 1 | 2 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3 | 2 | 6 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 1 | 2 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2 | 2 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 5 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1 | 2 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0 | 1 | 0
Flushing (Vascular disorders) | 3 | 0 | 1 | 2 | 0 | 0
Hypertension (Vascular disorders) | 5 | 2 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.